CLINICAL TRIAL: NCT07199478
Title: Application of an Intelligently Integrated Digital Rehabilitation Model Combining mHealth and ERAS in Total Hip and Knee Arthroplasty
Brief Title: Ntelligently Integrated Digital Rehabilitation Model Combining mHealth and ERAS in Total Hip and Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, XiaoYue Li, The Affiliated Hospital Of Southwest Medical University, The Affiliated Hospital Of Southwest Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH9H-2024-001
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty; Total Hip Arthroplasty; ERAS

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Participants received the standardized Enhanced Recovery After Surgery (ERAS) protocol plus the digital intervention via the "Joint Recovery Assistant" WeChat mini-program.
  Interventions: Procedure: Integrated mHealth and ERAS Digital Rehabilitation via WeChat Mini-Program
- Control group：Standardized ERAS Protocol (Placebo Comparator): Standardized ERAS Protocol
  Interventions: Procedure: Standardized ERAS Protocol

INTERVENTIONS:
Procedure: Integrated mHealth and ERAS Digital Rehabilitation via WeChat Mini-Program — This intervention arm is distinguished by the following key features:
  Theory-Driven Design: Uniquely integrates three established behavioral theories into its core functionality: Bandura's Self-Efficacy Theory, the Health Belief Model, and Illeris's Learning Model. This theoretical foundation directly informs the app's features to target psychological and behavioral barriers to recovery.
  Multi-Functional Platform: Combines several evidence-based components into a single, cohesive platform within the ubiquitous WeChat ecosystem. Key features include:
  Visual Goal and Progress Tracking: Provides patients with "mastery experiences."
  Peer Community ("Modeling Community"): Features patient stories and videos to provide "vicarious experiences" and social support.
  AI-Powered Persuasion System: Delivers automated, personalized feedback and remote encouragement from healthcare providers.
  Built-in Emotional Management Tools: Includes an emotion diary
  Other Names: Standardized ERAS Protocol
  Arms: Intervention Group
Procedure: Standardized ERAS Protocol — Participants received only the standardized Enhanced Recovery After Surgery (ERAS) protocol, representing the conventional care model.
  Arms: Control group：Standardized ERAS Protocol

SUMMARY:
Protocol

This study is a single-center, randomized controlled trial designed to evaluate the effectiveness of a WeChat-based mini-program mobile health (mHealth) intervention combined with an Enhanced Recovery After Surgery (ERAS) protocol for postoperative rehabilitation in patients undergoing total hip arthroplasty (THA) and total knee arthroplasty (TKA). The study will be conducted at the Affiliated Hospital of Southwest Medical University from July 2025 to December 2025, approved by the Ethics Committee (SH9H-2025-021), and registered on a clinical trials platform.

The study population consists of adults scheduled for unilateral primary THA or TKA, aged 18-80 years, with basic smartphone proficiency. Exclusion criteria include revision surgery, bilateral surgery, severe cognitive impairment, or baseline depression. Using a block randomization method stratified by surgical site (hip vs. knee), eligible participants will be allocated in a 1:1 ratio to either the intervention group (ERAS + "Joint Rehabilitation Assistant" mini-program) or the control group (ERAS only). The control group receives standard ERAS management, while the intervention group additionally uses the theoretically-grounded mini-program (based on self-efficacy theory, health belief model, and learning theory), which provides personalized rehabilitation plans, progress tracking, community interaction, and emotional support.

The primary outcome is physical function (HOOS-PS/KOOS-PS) at 6 weeks postoperatively. Secondary outcomes include pain, psychological status, quality of life, and safety indicators. The calculated sample size is 70 patients per group (total 140), accounting for a 20% dropout rate. Statistical analysis will follow the intention-to-treat principle, using linear mixed models to compare intergroup differences, with subgroup and sensitivity analyses performed. All outcome assessments will be conducted by blinded personnel to ensure data quality.

This protocol aims to validate the effectiveness and safety of the integrated digital rehabilitation model in improving functional recovery and quality of life, providing evidence-based support for post-arthroplasty rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old. Surgery Type: Scheduled to undergo unilateral primary total hip arthroplasty (THA) or total knee arthroplasty (TKA).

Physical Status: American Society of Anesthesiologists (ASA) classification I-III.

Digital Literacy: Confirmed ability to use a smartphone via a standardized digital literacy test.

Compliance: Willing and able to adhere to the study protocol.

Exclusion Criteria:

* Surgery Type: Revision surgery or simultaneous bilateral surgery. Cognitive Function: Presence of severe cognitive impairment (Mini-Mental State Examination (MMSE) score <24).

Arthritis Type: Inflammatory arthritis (e.g., rheumatoid arthritis). Psychological Status: Presence of depressive state at baseline (Hospital Anxiety and Depression Scale (HADS) depression subscale score ≥15).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Physical Function at 6 weeks post-surgery, measured by the Hip disability and Osteoarthritis Outcome Score-Physical Function Shortform (HOOS-PS) or Knee injury and Osteoarthritis Outcome Score-Physical Function Shortform (KOOS-PS) | 6 weeks post-surgery
  Standardized Video Interview: The outcome was assessed by blinded evaluators using a standardized video interview protocol to ensure consistency and reduce assessment bias, unlike studies using unblinded in-person assessments or unstandardized patient self-report.
  Joint-Specific Patient-Reported Outcome Measures (PROMs): Uses validated, joint-specific short forms (HOOS-PS/KOOS-PS) that are optimized for measuring physical function in the target population, rather than generic functional scales.
  Early Post-Discharge Timepoint: The primary endpoint is set at 6 weeks, a key early post-discharge period where digital intervention support is hypothesized to have the greatest impact on functional recovery trajectories, as opposed to longer-term endpoints (e.g., 6 months or 1 year).

SECONDARY OUTCOMES:
Pain Intensity | Baseline (preoperatively), 6 weeks, and 10 weeks postoperatively.
  Assessed using the Numerical Rating Scale (NRS, range 0-10) for pain at rest and during activity. A higher score indicates more severe pain.
Psychological Status | Baseline (preoperatively), 6 weeks, and 10 weeks postoperatively.
  Evaluated using the Hospital Anxiety and Depression Scale (HADS). This scale consists of two subscales for anxiety (HADS-A) and depression (HADS-D) to screen for emotional distress.
Self-Efficacy | Timepoints: Baseline (preoperatively), 6 weeks, and 10 weeks postoperatively.
  Assessed using the Self-Efficacy for Rehabilitation (SER) scale to measure patients' confidence in their ability to perform activities and tasks required for recovery.
Safety Outcomes | Timepoints: Monitored continuously from randomization until the 10-week follow-up visit.
  All adverse events (AEs) and serious adverse events (SAEs)-such as delayed wound healing, deep vein thrombosis, and infection-were recorded and compared between groups to evaluate the safety profile of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan, China

IPD SHARING:
Plan to Share IPD: No